CLINICAL TRIAL: NCT06219772
Title: Assessment of Dynamic Balance in Females With Adolescent Idiopathic Scoliosis Compared to Normal Subjects: A Comparative Study
Brief Title: Assessment of Dynamic Balance in Idiopathic Scoliosis Compared to Normal Subjects
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: King Khalid University (Other)
Responsible Party: Principal Investigator, Doaa Ayoub Elimy Mohammed, Lecturer of physical therapy for basic science department., faculty of physical Therapy, Cairo University
Other Study IDs: ECM#2023-2105
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Scoliosis
Keywords: adolescent idiopathic scoliosis; dynamic balance; Cobb angle; stability index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess dynamic balance in females with adolescent idiopathic scoliosis compared to normal subjects.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is one of the most common forms of scoliosis. It is a three-dimensional deformity of the spine and trunk with a lateral deviation of ≥ 10°, which can occur during the growing years from 10 years to puberty, with an apparent gender dominance rising with age and severity with a female to male ratio of 1.5:1 to 10:1.

Dynamic balance is the ability to maintain and regain the center of gravity within the base of support in response to outside perturbations or voluntary movements. It has been reported that AIS is associated with trunk imbalance and could negatively influence the sensorimotor control of posture and decrease postural balance capabilities, which increases susceptibility to injuries and impacts the individual's ability to engage in daily living activities.

Previous research reported that postural stability control in adolescents with idiopathic scoliosis is as good as in healthy individuals, and others found that AIS patients have poorer static balance control than age-matched patients without AIS. So the current study will be conducted to investigate the dynamic balance in females with adolescent idiopathic scoliosis compared to normal subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 10-20 years.
2. Idiopathic scoliosis will be diagnosed based on clinical examination and radiological measures.
3. Cobb's angle will be between 20° and 40°.
4. Their BMI from 18 to 24.9 kg/m2.
5. They must be willing to participate in the study.

Exclusion Criteria:

1. History of previous back surgery.
2. Neurological deficit.
3. Current lower extremity symptoms.
4. Symptoms of vertigo or dizziness.
5. No other disorders in the vertebral column (disc prolapse, spondylosis, fracture).

Ages: 10 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Adolescent idiopathic scoliosis and normal subjects
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | Through study completion, an average of 7 months
  A Biodex balance system will be used for measuring the dynamic balance.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada MR Koura, Ass. prof, Study Director — King Khalid University, Saudi Arabia
Locations (1):
- Doaa Ayoub Elimy, Cairo, Egypt